CLINICAL TRIAL: NCT07258927
Title: Comparison of the Effects of Integrated Neuromuscular Inhibition and Muscle Energy Techniques Combined With Core Stabilization Exercises in Patients With Chronic Mechanical Low Back Pain
Brief Title: Neuromuscular Inhibition vs Muscle Energy Techniques With Core Exercises in Mechanical Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melek Agırtmış, PT, PhD Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-GSHS-2025-INITKET-01
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Mechanical Low Back Pain
Keywords: Chronic mechanical low back pain; Integrated neuromuscular inhibition technique; Respiratory muscle strength; Core stabilization exercises; Muscle energy technique

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into three parallel groups:
  1. CSE + INIT
  2. CSE + MET
  3. CSE alone.
Who Masked: Outcomes Assessor
Masking Description: The investigator performing outcome assessments will be blinded to group allocation. Participants and care providers cannot be blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Stabilization + INIT (Experimental): Participants receive Core Stabilization Exercises (CSE) combined with Integrated Neuromuscular Inhibition Technique (INIT). Sessions are administered by a physiotherapist, 45-60 minutes per session, 3 times per week for 6 weeks. INIT includes ischemic compression, strain-counterstrain, and muscle energy techniques applied to active trigger points.
  Interventions: Behavioral: Core Stabilization Exercise (CSE); Behavioral: Integrated Neuromuscular Inhibition Technique (INIT)
- Core Stabilization + MET (Active Comparator): Participants receive Core Stabilization Exercises (CSE) combined with Muscle Energy Technique (MET) delivered by a physiotherapist, 45-60 minutes per session, 3 times per week for 6 weeks. Manual techniques target trigger points of quadratus lumborum, iliopsoas, hamstring, and erector spinae muscles.
  Interventions: Behavioral: Core Stabilization Exercise (CSE); Behavioral: Muscle Energy Technique (MET)
- Core Stabilization Only (Active Comparator): Participants perform only Core Stabilization Exercises (CSE), emphasizing activation of deep stabilizers (transversus abdominis and multifidus) with progressive exercises performed under physiotherapist supervision, 45-60 minutes per session, 3 times per week for 6 weeks.
  Interventions: Behavioral: Core Stabilization Exercise (CSE)

INTERVENTIONS:
Behavioral: Core Stabilization Exercise (CSE) — Supervised core stabilization exercise program focusing on activation of deep trunk stabilizers (transversus abdominis and multifidus). Training includes isolated activation, quadruped exercises, bridging variations, and functional stabilization drills. Sessions last 45-60 minutes, 3 times per week for 6 weeks and are delivered by a physiotherapist.
Behavioral: Integrated Neuromuscular Inhibition Technique (INIT) — Manual therapy combining ischemic compression, strain-counterstrain, and muscle energy techniques applied to active trigger points in the lumbar/pelvic region. Target muscles include quadratus lumborum, iliopsoas, hamstrings, and erector spinae. Sessions last 45-60 minutes with integrated exercise, 3 times per week for 6 weeks and are administered by a physiotherapist.
  Arms: Core Stabilization + INIT
Behavioral: Muscle Energy Technique (MET) — Manual technique using therapist-guided isometric contraction of shortened muscles followed by relaxation and passive stretch. Target muscles include quadratus lumborum, iliopsoas, hamstrings, and erector spinae. Sessions last 45-60 minutes with integrated exercise, 3 times per week for 6 weeks and are administered by a physiotherapist.
  Arms: Core Stabilization + MET

SUMMARY:
Chronic mechanical low back pain (CMLBP) is a common clinical problem that affects physical function, spinal mobility, and quality of life. Manual therapy techniques such as Integrated Neuromuscular Inhibition Technique (INIT) and Muscle Energy Technique (MET) are frequently used in clinical practice to reduce pain and improve function. Core stabilization exercises (CSE) have also been reported to enhance spinal stability and neuromuscular control. However, limited evidence exists comparing the combined effects of these manual therapy techniques with core stabilization exercise on clinical outcomes in individuals with CMLBP.

This randomized controlled clinical study aims to compare the effects of CSE combined with INIT and CSE combined with MET on pain intensity, functional disability, lumbar range of motion, psychosocial status, muscle endurance, and quality of life in adults with chronic mechanical low back pain.

Participants will be randomly assigned to one of two groups: (1) CSE + INIT or (2) CSE + MET. Each group will receive treatment two times per week for six weeks. Pain severity, functional status, lumbar mobility, patient-reported outcomes, and muscle endurance will be assessed at baseline, immediately after the intervention, and at follow-up.

The results of this study will help determine whether INIT or MET provides additional benefit when combined with core stabilization exercise for improving symptoms and function in individuals with chronic mechanical low back pain.

DETAILED DESCRIPTION:
Chronic mechanical low back pain (CMLBP) is one of the most prevalent musculoskeletal disorders worldwide. It is characterized by pain originating from the lumbar spine or surrounding structures without a specific underlying pathology. The condition often results in pain, functional disability, reduced spinal mobility, impaired muscle performance, and psychosocial effects, which can negatively influence quality of life.

Manual therapy modalities are commonly used in rehabilitation to alleviate symptoms and improve mobility in individuals with CMLBP. The Integrated Neuromuscular Inhibition Technique (INIT) is a multimodal approach that includes strain-counterstrain, trigger point release, and muscle energy technique to reduce muscle tension, deactivate tender points, and improve neuromuscular balance. Muscle Energy Technique (MET) is an osteopathic manual therapy approach that uses voluntary muscle contractions against resistance to relax hypertonic muscles, increase joint mobility, and reduce pain. Both techniques are frequently used in practice, yet their comparative effectiveness when combined with core stabilization exercise remains unclear.

Core Stabilization Exercises (CSE) focus on enhancing the strength, endurance, and motor control of the deep spinal stabilizing muscles. They are widely recommended to improve spinal stability, decrease pain, and enhance function in individuals with CMLBP.

This randomized controlled study aims to evaluate and compare the effectiveness of CSE combined with INIT versus CSE combined with MET on multiple clinical outcomes in individuals with CMLBP. Participants who meet the inclusion criteria will be randomly assigned to one of two intervention groups:

CSE + INIT Group: will receive integrated neuromuscular inhibition techniques along with core stabilization exercises.

CSE + MET Group: will receive muscle energy techniques along with core stabilization exercises.

Both groups will receive treatment twice weekly for six weeks. Outcome measures will include:

Pain intensity (e.g., Visual Analog Scale)

Functional disability (e.g., Oswestry Disability Index)

Lumbar range of motion

Muscle endurance

Psychosocial status

Quality of life

Assessments will be conducted at three time points: baseline, post-treatment, and follow-up.

The primary hypothesis is that both treatment approaches will lead to improvements in pain and function, but the combination of CSE with INIT may demonstrate superior outcomes compared to CSE with MET.

The findings of this study will provide valuable knowledge to clinicians regarding optimal manual therapy integration with exercise for individuals with chronic mechanical low back pain. This may contribute to evidence-based clinical decision-making and improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Diagnosed chronic mechanical low back pain (>3 months)
* Pain localized between T12 and gluteal fold
* Ability to follow exercise instructions
* Voluntary consent

Exclusion Criteria:

* Spine surgery history
* Herniated disc with neurological deficit
* Systemic neuromuscular or rheumatologic disease
* Acute lumbar trauma
* Pregnancy
* Current participation in another clinical trial
* Use of analgesics, muscle relaxants, or physiotherapy within the past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | Baseline, Week 6 (post-treatment)
  Pressure pain threshold will be assessed using a handheld pressure algometer at standardized lumbar paraspinal trigger point regions. PPT is defined as the minimum pressure that produces pain. Higher values indicate reduced pain sensitivity.
  Units of Measure: Kilograms per square centimeter (kg/cm²)

SECONDARY OUTCOMES:
Disability Level (Oswestry Disability Index) | Baseline, Week 6
  Functional disability will be measured using the Oswestry Disability Index (ODI). Scores range from 0-100%, with higher scores indicating greater disability.
  Outcome Measure: Disability Level (Oswestry Disability Index)
  Functional disability will be assessed using the Oswestry Disability Index (ODI). The ODI score ranges from 0 to 100 points, with higher scores indicating greater disability and lower scores indicating less disability.
  The ODI evaluates a participant's level of functional impairment due to low back pain, including activities such as:
  Pain intensity
  Personal care
  Lifting
  Walking
  Sitting
  Standing
  Sleeping
  Sex life Units of Measure: Percent (%)
  Social life
  Traveling

OTHER OUTCOMES:
Trunk Flexor Muscle Endurance | Baseline, Week 6
  Trunk flexor endurance will be evaluated using a standardized trunk flexor isometric hold test. Time (seconds) is recorded; longer duration indicates better endurance.
  Units of Measure: Seconds
Respiratory Muscle Strength | Baseline, 6 week
  Respiratory muscle strength will be assessed using a digital manometer measuring maximal inspiratory (MIP) and expiratory (MEP) pressures. Higher values indicate greater respiratory muscle strength.
  Units of Measure: cmH₂O
Modified Schober Test | Baseline, Week 6 (post-treatment)
  Lumbar flexion mobility will be assessed using the Modified Schober Test. A mark is placed on the lumbar spine and the distance change during maximal forward flexion is measured. Higher values indicate greater lumbar spine mobility.
  Units of Measure: Centimeters (cm)
Lumbar Range of Motion (ROM) | Baseline, Week 6 (post-treatment)
  Lumbar flexion, extension, lateral flexion will be measured using a digital inclinometer. Higher values indicate greater mobility. Units of Measure: Degrees

CONTACTS AND LOCATIONS:
Overall Officials: RÜSTEM MUSTAFAOĞLU, Study Director — Istanbul University-Cerrahpaşa - Graduate School of Health Sciences
Locations (1):
- Istanbul University-Cerrahpaşa, Graduate School / Doctoral Program, Istanbul, BAŞAKŞEHİR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: General study protocol and information, including Istanbul University Cerrahpaşa Ethics Committee approval and protocol details. — https://www.istanbul.edu.tr/
- See also: Official clinical trials registry providing general study information. — https://clinicaltrials.gov/
- See also: Istanbul University institutional resources and study-related documentation. — https://www.istanbul.edu.tr/